CLINICAL TRIAL: NCT01870726
Title: A Phase Ib/II, Multi-center, Open-label Study of INC280 in Combination With Buparlisib in Patients With Recurrent Glioblastoma
Brief Title: Safety and Efficacy of INC280 and Buparlisib (BKM120) in Patients With Recurrent Glioblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X2204; 2013-000699-14 (EudraCT Number)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: c-MET Inhibitor; PI3K Inhibitor, PTEN Mutations, Homozygous Del. of PTEN or PTEN Neg. by IHC, c-Met Ampli. by FISH, INC280, BKM120, Buparlisib; Recurrent GBM
Keywords: Glioblastoma multiforme (GBM), glioblastoma, Grade IV Astrocytoma, brain tumor, brain cancer, giant cell glioblastoma, gliosarcoma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — capmatinib; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase Ib (Experimental): To estimate the safe dose of the combination INC280 and buparlisib
  Interventions: Drug: INC280; Drug: Buparlisib
- Phase II (Experimental): To estimate anti-tumor efficacy of INC280 single agent and in combination with buparlisib
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: INC280 — Phase Ib: INC280 was given at the starting dose of 200mg capsules twice daily with escalation to higher strengths.
  Phase II: INC280 was given at the dose of 400mg (tablets) twice daily.
Drug: Buparlisib — Buparlisib was given at the starting dose of 50mg once daily with escalation to higher strengths.
  Other Names: BKM120
  Arms: Phase Ib

SUMMARY:
The study assessed the safety and the dose of the combination of INC280 and buparlisib (BKM120), as well as the anti-tumor activity of the combination, in patients with recurrent glioblastoma with PTEN mutations, homozygous deletion of PTEN or PTEN negative by IHC. In addition, the anti-tumor activity of INC280 single agent should have been assessed in patients with recurrent glioblastoma with c-Met alteration.

DETAILED DESCRIPTION:
This was a multi-center, open-label, phase Ib/II study. The aim of the phase Ib part was to estimate the MTD and/or to identify the recommended phase II dose (RP2D) for the combination of INC280 and buparlisib, followed by the phase II part to assess the clinical efficacy of INC280 single agent and in combination with buparlisib (BKM120), and to further assess the safety of the combination. In addition, a surgical arm should have started concurrently with the phase II part, to determine the PK/PD profile of the study drug combination in patients undergoing tumor resection for recurrent glioblastoma after 7 to 10-days treatment.

RP2D was not declared due to a lack of efficacy of the combination in the phase Ib stage, and phase II was continued with INC280 monotherapy only.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Histologically confirmed diagnosis of glioblastoma (after initial tumor resection or biopsy) with radiographic evidence of recurrent tumor per RANO criteria.
* Phase Ib: Documented evidence of PTEN mutations, homozygous deletion of PTEN or PTEN negative (H Score <10) by IHC confirmed by local or central assessment.
* Phase II: Documented evidence of c-Met amplification (GCN>5) (fusion transcripts or mutant c-Met may be eligible after discussion with Novartis) or PTEN mutations, homozygous deletion of PTEN or PTEN negative (H Score <10) by central assessment.
* Must have received the following treatment for glioblastoma:

  •Prior treatment with radiotherapy and temozolomide; Note: A maximum of two prior chemotherapy/antibody regimens (including bevacizumab or other direct VEFG/VEGFR inhibitors) for recurrent disease are permitted.
* Representative archival tumor sample from glioblastoma (formalin-fixed paraffine embedded tissue) must be available.
* ECOG performance status ≤ 2.
* Able to swallow and retain oral medication.
* Patients in the surgical arm only: patients with recurrent glioblastoma must be eligible for surgical resection as deemed by the site Investigator.

Exclusion Criteria:

* Prior or current treatment with a c-MET inhibitor or HGF-targeting therapy
* Prior treatment with a PI3K and/or mTOR inhibitors for glioblastoma or for pre-existing neoplasm transformed to glioblastoma (applicable for combination treatment arm only)
* Received radiation (including therapeutic radioisotopes such as strontium 89) therapy ≤ 3 months prior to the first dose of study treatment and have not recovered from side effects of such therapy (≤ Grade 1) prior to the first dose of study treatment, except for alopecia.
* Receiving treatment with medications that are known strong inhibitors or inducers of CYP3A, and cannot be discontinued 7 days prior to the start of the treatment and during the course of the study.
* Receiving treatment with medications that are known CYP3A, CYP1A2, CYP2C8, CYP2C9 or CYP2C19 substrates with narrow therapeutic index, and cannot be discontinued during the course of the study.
* Receiving treatment with long acting proton pump inhibitors, and cannot be discontinued 3 days prior to the start of INC280 treatment and during the course of the study.
* Currently receiving warfarin or other coumadin-derived anticoagulants for treatment, prophylaxis or otherwise.
* Currently receiving increasing or chronic treatment ( > 5 days) with corticosteroids (e.g. dexamethasone > 4 mg/day or other corticosteroids equivalent dose) or another immunosuppressive agent.
* History of acute or chronic pancreatitis or any risk factors that may increase the risk of pancreatitis.
* Active cardiac disease or a history of cardiac dysfunction.
* Impairment of gastrointestinal (GI) function or GI disease that might significantly alter the absorption of study drug
* Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders (defined according to DSM- IV).
* Anxiety ≥ CTCAE grade 3
* Any of the following baseline laboratory values:

  * Hemoglobin < 9 g/dL
  * Platelet count < 75 x 109/L
  * Absolute neutrophil count (ANC) < 1.0 x 109/L
  * INR > 1.5
  * Serum lipase > normal limits for the institution
  * Asymptomatic serum amylase > grade 2
  * Potassium, magnesium, and calcium (corrected for albumin) > normal limits for the institution
  * Total bilirubin > 1.5 x ULN
  * Serum creatinine >1.5 x ULN or creatinine clearance ≤ 45 mL/min
  * Alanine aminotransferase (AST) or aspartate aminotransferase (ALT) > 3.0 x ULN (or < 5.0 x ULN if liver metastases are present)
  * Fasting plasma glucose > 120mg/dL or > 6.7 mmol/L
  * HbA1c > 8%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01-09 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (5):
  - Dana Farber Cancer Institute SC, Boston, Massachusetts
  - Columbia University Medical Center- New York Presbyterian Dept of Oncology, New York, New York
  - Memorial Sloan Kettering Cancer Center Neurology, New York, New York
  - Duke University Medical Center Duke - Baker, Durham, North Carolina
  - University of Texas MD Anderson Cancer Center SC-3, Houston, Texas
- Germany (3):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Tübingen
- Netherlands (2):
  - ErasmusMC Cancer Institute - Neurooncology, RM G3-55, Rotterdam
  - University Medical Center Utrecht, Rm Q05.4.300, P.O. Box 85500, Utrecht
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] van den Bent M, Azaro A, De Vos F, Sepulveda J, Yung WKA, Wen PY, Lassman AB, Joerger M, Tabatabai G, Rodon J, Tiedt R, Zhao S, Kirsilae T, Cheng Y, Vicente S, Balbin OA, Zhang H, Wick W. A Phase Ib/II, open-label, multicenter study of INC280 (capmatinib) alone and in combination with buparlisib (BKM120) in adult patients with recurrent glioblastoma. J Neurooncol. 2020 Jan;146(1):79-89. doi: 10.1007/s11060-019-03337-2. Epub 2019 Nov 27. PMID 31776899

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 43 patients enrolled in this trial, 33 patients in the Phase Ib part of the study (patients were assigned to 6 dose combinations of INC280 with buparlisib) and 10 patients in the Phase II part of the study.
Groups:
- 200 mg BID Cap+50 mg QD: Phase Ib: The combination of 200mg INC280 (BID) capsule and 50 mg Buparlisib (QD) once daily for Phase Ib.
- 400 mg BID Cap+50 mg QD: Phase Ib: The combination of 400 mg INC280 (BID) capsule and 50mg Buparlisib (QD) once daily for Phase Ib.
- 500 mg BID Cap+50 mg QD: Phase Ib: The combination of 500 mg INC280 (BID) capsule and 50mg Buparlisib (QD) once daily for Phase Ib.
- 500 mg BID Cap+80 mg QD: Phase Ib: The combination of 500 mg INC280 (BID) capsule and 80mg Buparlisib (QD) once daily for Phase Ib.
- 300 mg BID Tab +80 mg QD: Phase Ib: The combination of 300 mg INC280 (BID) tablet and 80mg Buparlisib (QD) once daily for Phase Ib.
- 400 mg BID Tab +80 mg QD: Phase Ib: The combination of 400 mg INC280 (BID) tablet and 80mg Buparlisib (QD) once daily for Phase Ib.
- 400 mg BID Tab: Phase II: 400 mg INC280 (BID) tablet
Period: Overall Study
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab +80 mg QD | 400 mg BID Tab
Started | 5 | 6 | 4 | 6 | 7 | 5 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 4 | 6 | 7 | 5 | 10
Not completed — Withdrawal of informed consent | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Progressive disease | 5 | 5 | 4 | 5 | 6 | 4 | 10

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS comprised all patients who received at least one full or partial dose of study treatment. Patients were classified according to the planned treatment.
Groups:
- 500 mg BID Cap+80 mg QD: Phase Ib: The combination of 400 mg INC280 (BID) capsule and 80mg Buparlisib (QD) once daily for Phase Ib.
- Total: Total of all reporting groups
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab +80 mg QD | 400 mg BID Tab | Total
Number analyzed (Participants) | 5 | 6 | 4 | 6 | 7 | 5 | 10 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 4 | 5 | 4 | 4 | 10 | 35
  >=65 years | 3 | 0 | 0 | 1 | 3 | 1 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 3 | 0 | 2 | 7 | 16
  Male | 5 | 4 | 2 | 3 | 7 | 3 | 3 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Dose Limiting Toxicities (DLTs) in Cycle 1
Description: A DLT is defined as an adverse event or abnormal laboratory value where the relationship to study treatment cannot be ruled out, and is not primarily related to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle of treatment (28 days) with INC280 in combination with buparlisib and meets any of the pre-defined criteria. The maximum tolerated dose was identified as INC280 300 mg BID + buparlisib 80 mg QD.
Time Frame: Cycle 1, 28 days
Population: Dose determining set (DDS) consisted of all patients from the SAS who either met the minimum exposure criterion and had sufficient safety evaluations during Cycle 1, or discontinued earlier due to DLT during Cycle 1.
Measure: Number; unit: Number of Patients
Groups:
- 400 mg BID Tab+80 mg QD: Phase Ib: The combination of 400 mg INC280 (BID) tablet and 80mg Buparlisib (QD) once daily for Phase Ib.
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 4 | 5 | 4 | 6 | 7 | 4
Number of Patients
  Personality Change | 0 (1257.87) [1870.1 to 4978.4] | 1 (2291.80) [1010.1 to 5581.5] | 0 (2604.72) [1716.5 to 8086.8] | 0 (2702.56) [2463.8 to 8018.8] | 0 (2702.47) [1657.2 to 8924.7] | 0 (5627.79) [2978.3 to 13776.6]
  Nausea | 0 [4045.6 to 10405.8] | 0 [3069.8 to 13946.9] | 0 [6276.0 to 31532.5] | 0 [1940.8 to 3618.0] | 1 [8606.0 to 16381.0] | 0 [11576.1 to 17422.8]
  Aspartate Aminotransferase Increased | 0 [3880.4 to 7192.8] | 0 [2655.6 to 2655.6] | 0 [19903.7 to 27092.8] | 0 [4793.3 to 14289.7] | 0 [7002.3 to 12184.7] | 2 [13051.1 to 13051.1]

2. Primary Outcome: Phase II: Progression Free Survival Rate (PFSR)
Description: Estimated rate of patients treated during 6 months without experiencing disease progression.
  The Progression Free Survival Rate at 6 months was to be estimated using a Bayesian model described in the protocol. The models operating characteristics were evaluated based on the enrollment of at least 30 patients enrolled. Patients did not reach the milestone for the PFSR analysis (trial terminated); as such no analysis was performed.
Time Frame: 6 months
Population: Based on the phase I, a RP2D was not determined for the combination arm (Phase II combination arms were not opened). Patients did not reach the milestone needed for the PFSR analysis (at minimum the Bayesian model requires 30 patients) due to early termination, as such no analysis for PFSR was performed.
Groups:
- BID Tab+Buparlisib: Phase II: INC280 (BID) as a single agent and in combination with buparlisib
Arm/Group | BID Tab+Buparlisib
Number analyzed (Participants) | 0

3. Primary Outcome: Phase II Surgical Arm: Concentrations of INC280 and Buparlisib in Tumor.
Description: Concentrations of INC280 and buparlisib in tumor tissue.
Time Frame: 7 days
Population: Based on the phase I, a RP2D was not determined for the combination and the phase II combination arms were not opened.
Groups:
- BID + QD: The combination of INC280 (BID) and Buparlisib (QD).
Arm/Group | BID + QD
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Adverse Events
Description: To characterize the safety of INC280 single agent and in combination with buparlisib including type, frequency, severity of adverse events, serious adverse events, and dose interruptions and adjustments. Adverse events will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, unless otherwise specified.
  If CTCAE grading did not exist for an AE, the severity of mild, moderate, severe, and lifethreatening, corresponding to Grades 1 - 4, were used. CTCAE Grade 5 (death) was not used in this study but was collected as a seriousness criterion; rather, information about deaths was collected though a Death form.
Time Frame: throughout the duration of the trial, approximately 3 years from FPFV to LPLV
Population: Safety Analysis Set (SAS): The SAS comprised all patients who received at least one full or partial dose of study treatment. Patients were analyzed according to the treatment actually received. The SAS was used for all safety analyses.
Measure: Number; unit: Participants
Groups:
- 300 mg BID Tab + 80 mg QD: Phase Ib: The combination of 300 mg INC280 (BID) tablet and 80mg Buparlisib (QD) once daily for Phase Ib.
- 400 mg BID Tab + 80 mg QD: Phase Ib: the combination of 400 mg INC280 (BID) tablet and 80 mg Buparlisib (QD) once daily
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab + 80 mg QD | 400 mg BID Tab + 80 mg QD | 400 mg BID Tab
Number analyzed (Participants) | 5 | 6 | 4 | 6 | 7 | 5 | 9
Participants
  Adverse events | 5 | 6 | 4 | 6 | 7 | 5 | 9
  Treatment-related AEs | 4 | 4 | 4 | 4 | 7 | 5 | 6
  AEs with grade ≥ 3 | 5 | 4 | 4 | 2 | 5 | 4 | 8
  SAEs | 3 | 2 | 3 | 3 | 3 | 4 | 2
  AEs leading to discontinuation | 0 | 0 | 0 | 0 | 1 | 1 | 0
  AEs leading to dose adjustment/interruption | 2 | 3 | 2 | 4 | 4 | 4 | 5
  AEs requiring additional therapy | 4 | 5 | 3 | 5 | 7 | 5 | 7

5. Secondary Outcome: Pharmacokinetic Profile of INC280 - AUCtau
Description: Plasma concentration profile of INC280 in combination with Buparlisib. AUCtau is the AUC from time zero to the end of dosing interval.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, approximately 6 months
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all patients who provided an evaluable PK profile.
Measure: Median (Full Range); unit: hr*ng/ml
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 5 | 5 | 4 | 6 | 4 | 5
hr*ng/ml
  Cycle 1 Day 1 | 2435.6 (1257.87) [1870.1 to 4978.4] | 3005.9 (2291.80) [1010.1 to 5581.5] | 4789.7 (2604.72) [1716.5 to 8086.8] | 5071.7 (2702.56) [2463.8 to 8018.8] | 5732.2 (2702.47) [1657.2 to 8924.7] | 11127.7 (5627.79) [2978.3 to 13776.6]
  Cycle 1 Day 15 | 5749.3 [4045.6 to 10405.8] | 11261.7 [3069.8 to 13946.9] | 10581.0 [6276.0 to 31532.5] | 2779.4 [1940.8 to 3618.0] | 12801.3 [8606.0 to 16381.0] | 16590.6 [11576.1 to 17422.8]
  Cycle 2 Day 1 | 4894.6 [3880.4 to 7192.8] | 2655.6 [2655.6 to 2655.6] | 23498.3 [19903.7 to 27092.8] | 10554.3 [4793.3 to 14289.7] | 9593.5 [7002.3 to 12184.7] | 13051.1 [13051.1 to 13051.1]

6. Secondary Outcome: Pharmacokinetic Profile of INC280 - Cmax
Description: Plasma concentration profile of INC280 in combination with Buparlisib. Cmax is the Maximum (peak) observed drug concentration after dose administration.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, approximately 6 months
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all patients who provided an evaluable PK profile.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 5 | 5 | 4 | 6 | 4 | 5
ng/ml
  Cycle 1 Day 1 | 618.0 (509.47) [406.0 to 1680.0] | 880.0 (481.70) [219.0 to 1410.0] | 960.5 (898.05) [434.0 to 2510.0] | 860.0 (1081.12) [195.0 to 2770.0] | 1990.0 (778.91) [423.0 to 2510.0] | 3635.0 (1499.76) [1210.0 to 4640.0]
  Cycle 1 Day 15 | 1560.0 [745.0 to 2610.0] | 2005.0 [763.0 to 3930.0] | 3480.0 [1350.0 to 8350.0] | 545.5 [315.0 to 776.0] | 3610.0 [2320.0 to 4940.0] | 4850.0 [1800.0 to 5350.0]
  Cycle 2 Day 1 | 1200.0 [578.0 to 1540.0] | 2142.5 [675.0 to 3610.0] | 5010.0 [4230.0 to 5790.0] | 2254.5 [479.0 to 3740.0] | 3080.0 [2720.0 to 3440.0] | 3220.0 [3220.0 to 3220.0]

7. Secondary Outcome: Pharmacokinetic Profile of INC280 - Tmax
Description: Plasma concentration profile of INC280 in combination with Buparlisib. Tmax is the time to reach maximum (peak) observed concentration (Cmax) after dose administration
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, approximately 6 months
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all patients who provided an evaluable PK profile.
Measure: Median (Full Range); unit: hr
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 5 | 5 | 4 | 6 | 4 | 5
hr
  Cycle 1 Day 1 | 1.1 (509.47) [1.0 to 2.0] | 2.0 (481.70) [2.0 to 4.0] | 1.5 (898.05) [1.0 to 2.2] | 1.3 (1081.12) [1.1 to 4.0] | 1.6 (778.91) [1.0 to 2.2] | 2.0 (1499.76) [0.9 to 2.0]
  Cycle 1 Day 15 | 1.9 [0.9 to 2.0] | 2.0 [1.0 to 2.1] | 2.0 [1.0 to 2.1] | 2.6 [1.2 to 4.0] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.1]
  Cycle 2 Day 1 | 2.0 [1.0 to 4.0] | 2.0 [2.0 to 2.0] | 1.5 [1.0 to 2.1] | 2.1 [1.5 to 4.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0]

8. Secondary Outcome: Pharmacokinetic Profile of INC280 - T1/2
Description: Plasma concentration profile of INC280 in combination with Buparlisib. T1/2 is the terminal half life
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, approximately 6 months
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all patients who provided an evaluable PK profile.
Measure: Median (Full Range); unit: hr
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 5 | 5 | 4 | 6 | 4 | 5
hr
  Cycle 1 Day 15 | 13.4 [4.1 to 31.2] | 20.8 [16.3 to 28.6] | 26.0 [13.2 to 28.1] | 7.3 [7.3 to 7.3] | 13.1 [7.0 to 19.3] | 8.0 [4.2 to 28.0]
  Cycle 2 Day 1 | 9.9 [3.8 to 20.1] | 17.4 [17.4 to 17.4] | 26.3 [23.5 to 29.1] | 8.7 [5.8 to 11.5] | 6.3 [6.3 to 6.3] | 4.3 [4.3 to 4.3]

9. Secondary Outcome: Pharmacokinetic Profile of Buparlisib - AUCtau
Description: Plasma concentration profile of Buparlisib in combination with INC280. AUCtau is the AUC from time zero to the end of dosing interval.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, approximately 6 months
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all patients who provided an evaluable PK profile.
Measure: Median (Full Range); unit: hr*ng/ml
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 5 | 5 | 4 | 6 | 4 | 5
hr*ng/ml
  Cycle 1 Day 1 | 3072.0 (1257.87) [2119.7 to 3448.0] | 1865.0 (2291.80) [1383.2 to 3840.8] | 3328.2 (2604.72) [2830.2 to 4104.1] | 3825.8 (2702.56) [2784.0 to 5201.4] | 4425.3 (2702.47) [3109.8 to 5238.2] | 3658.8 (5627.79) [3347.7 to 5509.4]
  Cycle 1 Day 15 | 8728.5 [4874.3 to 10962.7] | 4591.9 [3167.1 to 10562.3] | 6108.4 [5300.5 to 7605.5] | 10844.6 [6761.7 to 14927.4] | 10366.5 [8257.8 to 11052.6] | 8535.1 [4102.2 to 8908.3]
  Cycle 2 Day 1 | 7930.8 [3563.5 to 9712.2] | 3776.7 [3477.6 to 4075.7] | 6976.0 [3436.1 to 10515.9] | 5903.0 [4850.4 to 12072.9] | 7857.2 [7757.7 to 9361.9] | 7344.3 [7344.3 to 7344.3]

10. Secondary Outcome: Pharmacokinetic Profile of Buparlisib - Cmax
Description: as for outcome 6
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, approximately 6 months
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all patients who provided an evaluable PK profile.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 5 | 5 | 4 | 6 | 4 | 5
ng/ml
  Cycle 1 Day 1 | 484.0 (509.47) [234.0 to 590.0] | 351.0 (481.70) [162.0 to 488.0] | 399.0 (898.05) [347.0 to 469.0] | 522.0 (1081.12) [333.0 to 776.0] | 508.0 (778.91) [373.0 to 711.0] | 475.0 (1499.76) [361.0 to 542.0]
  Cycle 1 Day 15 | 664.0 [568.0 to 791.0] | 459.0 [294.0 to 623.0] | 542.0 [456.0 to 791.0] | 785.0 [684.0 to 886.0] | 814.0 [628.0 to 1330.0] | 788.5 [390.0 to 1700.0]
  Cycle 2 Day 1 | 560.0 [290.0 to 813.0] | 377.5 [285.0 to 470.0] | 611.0 [409.0 to 813.0] | 529.5 [383.0 to 865.0] | 735.0 [558.0 to 890.0] | 600.0 [600.0 to 600.0]

11. Secondary Outcome: Pharmacokinetic Profile of Buparlisib - Tmax
Description: as for outcome 7
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, approximately 6 months
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all patients who provided an evaluable PK profile.
Measure: Median (Full Range); unit: hr
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 5 | 5 | 4 | 6 | 4 | 5
hr
  Cycle 1 Day 1 | 1.0 (509.47) [0.6 to 1.2] | 1.0 (481.70) [0.6 to 2.0] | 1.0 (898.05) [0.5 to 1.2] | 0.6 (1081.12) [0.5 to 2.0] | 1.2 (778.91) [0.5 to 2.0] | 1.0 (1499.76) [0.9 to 2.0]
  Cycle 1 Day 15 | 0.9 [0.9 to 1.0] | 2.0 [1.0 to 2.1] | 1.0 [1.0 to 2.0] | 1.6 [1.2 to 2.0] | 1.0 [0.5 to 1.0] | 1.3 [0.5 to 2.1]
  Cycle 2 Day 1 | 1.0 [0.5 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.8 [1.0 to 2.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

12. Secondary Outcome: Pharmacokinetic Profile of Buparlisib - T1/2
Description: Plasma concentration profile of INC280 in combination with Buparlisib. T1/2 is the terminal half life
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, approximately 6 months
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all patients who provided an evaluable PK profile.
Measure: Median (Full Range); unit: hr
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD
Number analyzed (Participants) | 5 | 5 | 4 | 6 | 4 | 5
hr
  Cycle 1 Day 15 | 37.3 [29.1 to 52.4] | 31.1 [18.7 to 46.4] | 21.8 [20.8 to 29.4] | 30.9 [19.9 to 41.8] | 38.0 [21.3 to 44.9] | 22.8 [5.8 to 31.5]
  Cycle 2 Day 1 | 34.0 [10.4 to 37.9] | 21.3 [16.4 to 26.1] | 27.0 [9.6 to 44.3] | 17.2 [16.8 to 31.9] | 20.1 [19.4 to 41.2] | 12.0 [12.0 to 12.0]

13. Secondary Outcome: Best Overall Response (BOR)
Description: Best Overall Response (BOR) observed in the study population of INC280 Single Agent and in Combination with Buparlisib. Responses will be assessed by the investigators following the RANO criteria with MRI or CT scans scheduled every 8 weeks.
  Summary of the RANO response criteria: CR has no T1-Gd+ (enhancing lesion), stable or decrease T2/FLAIR (non-enhancing lesion), absence of new lesion, stable or improve in clinical status; PR has ≥50% decrease T1-Gd+ (enhancing lesion), stable or decrease T2/FLAIR (non-enhancing lesion), absence of new lesion, stable or improve in clinical status; SD has ≥50% decrease but <25% increase T1-Gd+ (enhancing lesion), stable or decrease T2/FLAIR (non-enhancing lesion), absence of new lesion, stable or improve in clinical status; PD has ≥25% increase in T1-Gd+ (enhancing lesion), increase T2/FLAIR (non-enhancing lesion), presence of new lesion, deterioration in clinical status.
Time Frame: throughout the duration of the trial - approximately 3 years (from FPFV to LPLV)
Population: FAS
Measure: Number; unit: Participants
Groups:
- 400 mg BID Tab+80 mg QD: Phase Ib: The combination of 400 mg INC280 (BID) capsule and 80mg Buparlisib (QD) once daily for Phase Ib.
Arm/Group | 200 mg BID Cap+50 mg QD | 400 mg BID Cap+50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab +80 mg QD | 400 mg BID Tab+80 mg QD | 400 mg BID Tab
Number analyzed (Participants) | 5 | 6 | 4 | 6 | 7 | 5 | 10
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease (SD) | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Progressive Disease (PD) | 5 | 5 | 4 | 4 | 7 | 4 | 6
  Unknown (UNK) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Assessed | 0 | 1 | 0 | 1 | 0 | 1 | 1

14. Secondary Outcome: Overall Survival (OS)
Description: Survival rate of patients from start of treatment to date of death due to any cause.
  Patients did not reach the milestone for the survival data analysis (terminated early); as such no analysis was done.
Time Frame: throughout the duration of the trial - approximately 3 years (FPFV to LPLV)
Population: Based on the phase I, a RP2D was not determined for the combination arm (Phase II combination arms were not opened). Patients did not reach the milestone needed for the OS analysis (at minimum the Bayesian model requires 30 patients) due to early termination, as such no analysis for OS was done.
Groups:
- All Patients: The combination of INC280 (BID) and Buparlisib (QD).
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit, approximately 3 years.
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- INC280 200 mg BID Tab: Phase II: 200mg INC280 (BID) tablet in Phase II. A patient never received the intended PhII dose as planned (400 mg BID) but is resented as a separate group for safety.
- 400 mg BID Cap + 50 mg QD: Phase Ib: The combination of 400mg INC280 (BID) capsule and 50 mg Buparlisib (QD) once daily for Phase Ib.
- 500 mg BID Cap+50 mg QD: Phase Ib: The combination of 500mg INC280 (BID) capsule and 50 mg Buparlisib (QD) once daily for Phase Ib.
- 500 mg BID Cap+80 mg QD: Phase Ib: The combination of 500mg INC280 (BID) capsule and 80 mg Buparlisib (QD) once daily for Phase Ib.
- 300 mg BID Tab+ 80 mg QD: Phase Ib: The combination of 300mg INC280 (BID) capsule and 80 mg Buparlisib (QD) once daily for Phase Ib.
- 400 mg BID Tab+80 mg QD: Phase Ib: The combination of 400mg INC280 (BID) capsule and 80 mg Buparlisib (QD) once daily for Phase Ib.
- All Patients (Phase Ib): Phase Ib: All Patients with the combination of INC280 (BID) and Buparlisib (QD) once daily.
- 400 mg BID Tab: Phase II: 400mg INC280 (BID) tablet in Phase II.
- All Patients (Phase II): Phase II: All patients treated with INC280 (BID) tablet once daily in the Phase II.
Arm/Group | INC280 200 mg BID Tab | 200 mg BID Cap+50 mg QD | 400 mg BID Cap + 50 mg QD | 500 mg BID Cap+50 mg QD | 500 mg BID Cap+80 mg QD | 300 mg BID Tab+ 80 mg QD | 400 mg BID Tab+80 mg QD | All Patients (Phase Ib) | 400 mg BID Tab | All Patients (Phase II)
Serious Adverse Events (participants affected / at risk) | 1/1 | 3/5 | 2/6 | 3/4 | 3/6 | 3/7 | 4/5 | 18/33 | 2/9 | 3/10
Other Adverse Events (participants affected / at risk) | 0/1 | 5/5 | 6/6 | 4/4 | 6/6 | 7/7 | 5/5 | 33/33 | 9/9 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INC280 200 mg BID Tab (N=1) | 200 mg BID Cap+50 mg QD (N=5) | 400 mg BID Cap + 50 mg QD (N=6) | 500 mg BID Cap+50 mg QD (N=4) | 500 mg BID Cap+80 mg QD (N=6) | 300 mg BID Tab+ 80 mg QD (N=7) | 400 mg BID Tab+80 mg QD (N=5) | All Patients (Phase Ib) (N=33) | 400 mg BID Tab (N=9) | All Patients (Phase II) (N=10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
FEBRILE INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
PERITONITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ATAXIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0
BRAIN OEDEMA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PARAPARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
PARTIAL SEIZURES (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
SEIZURE (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 0
APATHY (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
EMBOLISM (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INC280 200 mg BID Tab (N=1) | 200 mg BID Cap+50 mg QD (N=5) | 400 mg BID Cap + 50 mg QD (N=6) | 500 mg BID Cap+50 mg QD (N=4) | 500 mg BID Cap+80 mg QD (N=6) | 300 mg BID Tab+ 80 mg QD (N=7) | 400 mg BID Tab+80 mg QD (N=5) | All Patients (Phase Ib) (N=33) | 400 mg BID Tab (N=9) | All Patients (Phase II) (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
DIPLOPIA (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 5 | 3 | 3
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 7 | 1 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 6 | 1 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 3 | 2 | 10 | 2 | 2
RECTAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 5 | 1 | 1
ASTHENIA (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1
CHILLS (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
FATIGUE (General disorders) | 0 | 2 | 3 | 1 | 2 | 2 | 2 | 12 | 3 | 3
GAIT DISTURBANCE (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4 | 1 | 1
PYREXIA (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
ORCHITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 2 | 2
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 1 | 1 | 0 | 2 | 4 | 9 | 0 | 0
AMYLASE INCREASED (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 1 | 1 | 0 | 2 | 3 | 8 | 0 | 0
BLOOD ALBUMIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 5 | 1 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 5 | 1 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GLOMERULAR FILTRATION RATE DECREASED (Investigations) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 0
INSULIN C-PEPTIDE INCREASED (Investigations) | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 6 | 0 | 0
LIPASE INCREASED (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 4 | 3 | 3
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0
PROTEIN TOTAL DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
PROTHROMBIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
WEIGHT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 6 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 1 | 2 | 0 | 7 | 1 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 4 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
AMNESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 0
ATAXIA (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
BRAIN OEDEMA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 7 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
DYSARTHRIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0
DYSKINESIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DYSMETRIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
EPILEPSY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
FACIAL PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
FACIAL PARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 2 | 0 | 1 | 2 | 2 | 2 | 9 | 4 | 4
HEMIANOPIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
HEMIANOPIA HOMONYMOUS (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 5 | 1 | 1
HEMIPLEGIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
LETHARGY (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 7 | 0 | 0
NEUROLOGIC NEGLECT SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
PARAPARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
PARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1
PYRAMIDAL TRACT SYNDROME (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SEIZURE (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 4 | 1 | 1
TREMOR (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VITH NERVE PARALYSIS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 6 | 1 | 1
APATHY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
BRADYPHRENIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
DEPRESSION (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 3 | 2 | 8 | 1 | 1
DISORIENTATION (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1
IRRITABILITY (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MOOD ALTERED (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
PERSONALITY CHANGE (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SLEEP DISORDER (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 2
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
SKIN ATROPHY (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
EMBOLISM (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1
HYPOTENSION (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
At the end of Phase Ib, it was decided not to enroll patients in the two Phase II arms evaluating INC280 with buparlisib. The phase II INC280 single agent arm was halted before it reached target enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.